CLINICAL TRIAL: NCT03083899
Title: DiaTast - Patient Reported Experience in a New Out-patient Structure With Patient-initiated Visits
Brief Title: The Diabetes Patient Takes Responsibility
Acronym: DiaTast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Claus Bogh Juhl, MD, PhD, Ass Professor, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Diatast
Record Dates: First submitted 2017-03-03; First posted 2017-03-20 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 1; Patient Reported Outcome; Health Care Economics and Organizations
Keywords: Diabetes; Organization; Out-patient control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diatast (Experimental): Free patient-initiated use of out-patient services
  Interventions: Other: Out-patient clinic on demand (patient-initiated)
- Control (Placebo Comparator): Scheduled diabetes control
  Interventions: Other: Scheduled out-patient clinic

INTERVENTIONS:
Other: Out-patient clinic on demand (patient-initiated) — Free use of any resources in the out-patient clinic
  Arms: Diatast
Other: Scheduled out-patient clinic — Scheduled use of the out-patient clinic
  Arms: Control

SUMMARY:
People with Type 1 diabetes (T1D) are randomized to follow the normal scheduled visit procedure in the outpatient clinic OR to have open access to the clinic, i.e. they can get an appointment with a nurse or doctor within defined time intervals via telephone, e-mail or apps. Patient-reported outcomes (patient satisfaction and experience, QoL) clinical variables (HbA1c, blood pressure etc.) and use of human resources (doctors, diabetes-nurses and diet physicians) are monitored.

DETAILED DESCRIPTION:
This is a 24 month prospective randomized controlled trial. People with Type 1 diabetes (T1D) are randomized to two groups: (i) Patients randomized to the control group receive their standard diabetes care and are seen in the out-patient clinic with regular intervals (typically a diabetes nurse every 3-4 month and a diabetes doctor once a year. (ii) Patients randomized to the intervention group are not called for at fixed time points. They can arrange visits in the diabetes clinic whenever they feel the need to do so. The have a guarantee for a consultation with a diabetes nurse within one week and with a diabetes doctor or diet physician within two weeks. Questionnaires (a specific questionnaire focused on patient satisfaction developed for the study and AddQoL) are filled in at time 0 and 24 month. Blood samples for diabetes-related variables (HbA1c, lipid status), blood pressure, body weight etc. are likewise recorded at time 0 and 24 month. Economic and time requirements are evaluated at 24 month.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetes 18 - 80 years Multiple injections or Insulin pump therapy

Exclusion Criteria:

Newly diagnosed T1D Psychiatric illness Need for translation Unstable conditions such as progressive retinopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome | 24 month
  Questionnaire regarding satisfaction of the out-patient clinic

SECONDARY OUTCOMES:
Clinical diabetes variables 1 | 24 month
  HbA1c
Health Care Economy | 24 month
  Use of resources in the out-patient clinic
Clinical diabetes variables 2 | 24 month
  Blood pressure
Clinical diabetes variables 3 | 24 month
  Lipids
Diabetes Dependent quality of Life | 24 month
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Juhl, MD PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of South West Jutland, University hospital of Southern Denmark, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No